CLINICAL TRIAL: NCT00460603
Title: A Randomized Phase 2 Study Of The Anti-Angiogenesis Agent AG-013736 In Combinations With Chemotherapy And Bevacizumab In Patients With Metastatic Colorectal Cancer Preceded By A Phase 1 Portion
Brief Title: Study With AG-013736 Combined With Chemotherapy And Bevacizumab In Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4061020
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Results first posted 2013-06-04 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-11

CONDITIONS: Colorectal Neoplasms
Keywords: GI neoplasms (phase 1)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- B (Active Comparator): bevacizumab 5 mg/kg every 2 weeks + FOLFOX
  Interventions: Drug: bevacizumab
- C (Experimental): AG-013726 5 mg bid+ bevacizumab 2 mg/kg every 2 weeks + FOLFOX
  Interventions: Drug: AG-013726
- A (Experimental): AG-013736 5 mg bid starting dose + FOLFOX
  Interventions: Drug: AG-013736 (axitinib)

INTERVENTIONS:
Drug: bevacizumab — bevacizumab 5 mg/kg every 2 weeks
  Arms: B
Drug: AG-013726 — AG-013726 5 mg bid every 2 weeks
  Arms: C
Drug: AG-013736 (axitinib) — AG-013736 5 mg bid starting dose
  Arms: A

SUMMARY:
To determine the safety and efficacy of AG-013736 in combination with other standard of care medication in patients with first line metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* (Phase 1) Patients with any solid/GI tumor who have had no more than 1 previous chemotherapy for greater than 3 months prior to enrollment
* (Phase 2) Patients with locally advanced or metastatic colorectal cancer (CRC) previously untreated with any systemic therapy.
* Patients treated with adjuvant chemotherapy (with radiation) will be eligible if last treatment was > 12 months prior to enrollment,
* Patients must have measurable disease by RECIST and if any history of hypertension, it must be controlled with medication.

Exclusion Criteria:

* Prior system therapy for advanced CRC (Ph 2 portion only)
* Prior treatment with anti-angiogenesis agent such as bevacizumab or VEGF inhibitors.
* Prior irradiation of greater than 25% of bone marrow (whole pelvis = 25%)
* Prior radiation, major surgery, or investigational agent within 4 weeks of study entry except palliative radiotherapy to non-target, metastatic lesions. Minor surgeries should be completed > 2 weeks of enrollment and be fully recovered from any procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2006-01; Primary Completion 2012-04 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (86):
- United States (86):
  - Pfizer Investigational Site, Daphne, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Antioch, California
  - Pfizer Investigational Site, Colton, California
  - Pfizer Investigational Site, Corona, California
  - Pfizer Investigational Site, Gilroy, California
  - Pfizer Investigational Site, Glendora, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Pleasant Hill, California
  - Pfizer Investigational Site, Pomona, California
  - Pfizer Investigational Site, Rancho Cucamonga, California
  - Pfizer Investigational Site, Rancho Mirage, California
  - Pfizer Investigational Site, Redlands, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Leandro, California
  - Pfizer Investigational Site, West Covina, California
  - Pfizer Investigational Site, Auroa, Colorado
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Lakewood, Colorado
  - Pfizer Investigational Site, Littleton, Colorado
  - Pfizer Investigational Site, Lone Tree, Colorado
  - Pfizer Investigational Site, Longmont, Colorado
  - Pfizer Investigational Site, Parker, Colorado
  - Pfizer Investigational Site, Thornton, Colorado
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Stuart, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Beech Grove, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Jeffersonville, Indiana
  - Pfizer Investigational Site, Muncie, Indiana
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Shelbyville, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Brownstone, Michigan
  - Pfizer Investigational Site, Dearborn, Michigan
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, West Bloomfield, Michigan
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Lee's Summit, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Grand Island, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Summit, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Amsterdam, New York
  - Pfizer Investigational Site, Hudson, New York
  - Pfizer Investigational Site, Latham, New York
  - Pfizer Investigational Site, Rexford, New York
  - Pfizer Investigational Site, Troy, New York
  - Pfizer Investigational Site, Kernersville, North Carolina
  - Pfizer Investigational Site, Lexington, North Carolina
  - Pfizer Investigational Site, Mount Airy, North Carolina
  - Pfizer Investigational Site, North Wilkesboro, North Carolina
  - Pfizer Investigational Site, Pollocksville, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Oregon City, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Tualatin, Oregon
  - Pfizer Investigational Site, West Reading, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Easley, South Carolina
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Seneca, South Carolina
  - Pfizer Investigational Site, Spartanburg, South Carolina
  - Pfizer Investigational Site, Chattanooga, Tennessee
  - Pfizer Investigational Site, Franklin, Tennessee
  - Pfizer Investigational Site, Gallatin, Tennessee
  - Pfizer Investigational Site, Hermitage, Tennessee
  - Pfizer Investigational Site, Lebanon, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Smyrna, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Tyler, Texas
  - Pfizer Investigational Site, Ogden, Utah
  - Pfizer Investigational Site, Everett, Washington
  - Pfizer Investigational Site, Kennewick, Washington
  - Pfizer Investigational Site, Vancouver, Washington

REFERENCES:
- [Derived] Hoh CK, Burris HA 3rd, Bendell JC, Tarazi J, Rosbrook B, Kim S, Infante JR, Reid TR. Intermittent dosing of axitinib combined with chemotherapy is supported by (18)FLT-PET in gastrointestinal tumours. Br J Cancer. 2014 Feb 18;110(4):875-81. doi: 10.1038/bjc.2013.806. Epub 2014 Jan 14. PMID 24423921
- [Derived] Infante JR, Reid TR, Cohn AL, Edenfield WJ, Cescon TP, Hamm JT, Malik IA, Rado TA, McGee PJ, Richards DA, Tarazi J, Rosbrook B, Kim S, Cartwright TH. Axitinib and/or bevacizumab with modified FOLFOX-6 as first-line therapy for metastatic colorectal cancer: a randomized phase 2 study. Cancer. 2013 Jul 15;119(14):2555-63. doi: 10.1002/cncr.28112. Epub 2013 Apr 19. PMID 23605883
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061020&StudyName=Study%20With%20AG-013736%20Combined%20With%20Chemotherapy%20And%20Bevacizumab%20In%20Patients%20With%20Metastatic%20Colorectal%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1): Bevacizumab 1 milligram per kilogram (mg/kg) intravenous infusion over 90 minutes on Day 1 of each 14-day cycle followed by FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 milligram per square meter (mg/m^2) intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently with oxaliplatin, then 5-fluorouracil (5-FU) 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily starting from Day 3 in Cycle 1 and starting from Day 1 in all subsequent cycles administered following bevacizumab infusion on Day 1. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 2): Bevacizumab 2 mg/kg intravenous infusion over 90 minutes on Day 1 of each 14-day cycle followed by FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently with oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily starting from Day 3 in Cycle 1 and starting from Day 1 in all subsequent cycles administered following bevacizumab infusion on Day 1. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 3): Bevacizumab 5 mg/kg intravenous infusion over 90 minutes on Day 1 of each 14-day cycle followed by FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently with oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily starting from Day 3 in Cycle 1 and starting from Day 1 in all subsequent cycles administered following bevacizumab infusion on Day 1. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 1: Axitinib + FOLFIRI (Cohort 4): FOLFIRI combination chemotherapy on Day 1 of each 14-day cycle consisting of irinotecan 180 mg/m^2 intravenous infusion over 90 minutes, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently with irinotecan, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily starting from Day 3 in Cycle 1 and starting from Day 1 in all subsequent cycles administered prior to irinotecan infusion on Day 1. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 1: Axitinib + FOLFOX (Cohort 5): FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently with oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily starting from Day 3 in Cycle 1 and starting from Day 1 in all subsequent cycles administered prior to oxaliplatin infusion on Day 1. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 1: Axitinib + FOLFIRI (Cohort 6): FOLFIRI combination chemotherapy on Day 1 of each 14-day cycle consisting of irinotecan 180 mg/m^2 intravenous infusion over 90 minutes, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently with irinotecan, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily from Day 3 to Day 12 in each 14-day cycle administered following completion of 5-FU infusion on Day 3. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 1: Axitinib + FOLFOX (Cohort 7): FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently with oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily starting from Day 3 to Day 12 in each 14-day cycle administered following completion of 5-FU infusion on Day 3. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 1: Axitinib + FOLFIRI (Cohort 8): Axitinib (AG-13736) tablet 7 mg orally twice daily for 7 days in 2-week lead-in period prior to Day 1 Cycle 1. FOLFIRI combination chemotherapy on Day 1 of each 14-day cycle consisting of irinotecan 180 mg/m^2 intravenous infusion over 90 minutes, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently with irinotecan, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 7 mg to 10 mg orally twice daily from Day 3 to Day 9 in each 14-day cycle administered following completion of 5-FU infusion on Day 3. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 1: Axitinib + FOLFIRI (Cohort 9): Axitinib (AG-13736) tablet 7 mg orally twice daily for 7 days in 2-week lead-in period prior to Day 1 Cycle 1. FOLFIRI combination chemotherapy on Day 1 of each 14-day cycle consisting of irinotecan 180 mg/m^2 intravenous infusion over 90 minutes, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently with irinotecan, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 10 mg orally twice daily from Day 3 to Day 9 in each 14-day cycle administered following completion of 5-FU infusion on Day 3. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 2: Axitinib + FOLFOX: FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently with oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily in each 14-day cycle administered prior to oxaliplatin infusion on Day 1. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 2: Bevacizumab + FOLFOX: Bevacizumab 5 mg/kg intravenous infusion over 90 minutes on Day 1 of each 14-day cycle followed by FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently with oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 2: Axitinib + Bevacizumab + FOLFOX: Bevacizumab 2 mg/kg intravenous infusion over 90 minutes on Day 1 of each 14-day cycle followed by FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently with oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily in each 14-day cycle administered following bevacizumab infusion on Day 1. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
Period: Phase 1
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1) | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 2) | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 3) | Phase 1: Axitinib + FOLFIRI (Cohort 4) | Phase 1: Axitinib + FOLFOX (Cohort 5) | Phase 1: Axitinib + FOLFIRI (Cohort 6) | Phase 1: Axitinib + FOLFOX (Cohort 7) | Phase 1: Axitinib + FOLFIRI (Cohort 8) | Phase 1: Axitinib + FOLFIRI (Cohort 9) | Phase 2: Axitinib + FOLFOX | Phase 2: Bevacizumab + FOLFOX | Phase 2: Axitinib + Bevacizumab + FOLFOX
Started | 6 | 6 | 4 | 8 | 6 | 4 | 6 | 3 | 18 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 4 | 8 | 6 | 4 | 6 | 3 | 18 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 1 | 1 | 2 | 0 | 0 | 3 | 0 | 4 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 1 | 2 | 2 | 2 | 2 | 2 | 11 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 1 | 3 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Other | 0 | 3 | 1 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1) | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 2) | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 3) | Phase 1: Axitinib + FOLFIRI (Cohort 4) | Phase 1: Axitinib + FOLFOX (Cohort 5) | Phase 1: Axitinib + FOLFIRI (Cohort 6) | Phase 1: Axitinib + FOLFOX (Cohort 7) | Phase 1: Axitinib + FOLFIRI (Cohort 8) | Phase 1: Axitinib + FOLFIRI (Cohort 9) | Phase 2: Axitinib + FOLFOX | Phase 2: Bevacizumab + FOLFOX | Phase 2: Axitinib + Bevacizumab + FOLFOX
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 42 | 43 | 41
Treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 39 | 43 | 41
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 42 | 43 | 41
Not completed — Ongoing in study A4061008 (NCT00828919) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 9 | 10
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 16 | 7
Not completed — Objective Progression or Relapse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 10 | 17
Not completed — Global Deterioration of Health Status | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 5
Not completed — Randomized, but not treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1): Bevacizumab 1 mg/kg intravenous infusion over 90 minutes on Day 1 of each 14-day cycle followed by FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently with oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily starting from Day 3 in Cycle 1 and starting from Day 1 in all subsequent cycles administered following bevacizumab infusion on Day 1. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1) | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 2) | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 3) | Phase 1: Axitinib + FOLFIRI (Cohort 4) | Phase 1: Axitinib + FOLFOX (Cohort 5) | Phase 1: Axitinib + FOLFIRI (Cohort 6) | Phase 1: Axitinib + FOLFOX (Cohort 7) | Phase 1: Axitinib + FOLFIRI (Cohort 8) | Phase 1: Axitinib + FOLFIRI (Cohort 9) | Phase 2: Axitinib + FOLFOX | Phase 2: Bevacizumab + FOLFOX | Phase 2: Axitinib + Bevacizumab + FOLFOX | Total
Number analyzed (Participants) | 6 | 6 | 4 | 8 | 6 | 4 | 6 | 3 | 18 | 42 | 43 | 41 | 187
Age, Customized [Number; unit: Participants]
  Less than (<) 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18 to 44 years | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 4 | 8 | 21
  45 to 64 years | 2 | 1 | 3 | 3 | 2 | 1 | 5 | 3 | 13 | 22 | 18 | 23 | 96
  Greater than or equal to (>=) 65 years | 3 | 3 | 1 | 4 | 3 | 2 | 1 | 0 | 4 | 18 | 21 | 10 | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 2 | 1 | 2 | 2 | 0 | 7 | 17 | 15 | 15 | 67
  Male | 3 | 5 | 2 | 6 | 5 | 2 | 4 | 3 | 11 | 25 | 28 | 26 | 120

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response: Phase 2
Description: Percentage of participants with objective response (OR) based assessment of confirmed complete response(CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed CR defined as disappearance of all lesions and no appearance of new lesions. Confirmed PR defined as >=30 percent (%) decrease in sum of the longest dimensions (LD) of the target lesions taking as reference the baseline sum LD , without progression of nontarget lesions and no appearance of new lesions. Confirmed responses are those that persist on repeat imaging study >=4 weeks after initial documentation of response.
Time Frame: Baseline (Phase 2) until disease progression, assessed every 6 weeks up to Week 148 (Phase 2) or follow-up (every 6 weeks after last dose of study drug until progression or start of alternate therapy)
Population: Intent-to-treat (ITT) population included all randomized participants, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug from that to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2: Axitinib + FOLFOX | Phase 2: Bevacizumab + FOLFOX | Phase 2: Axitinib + Bevacizumab + FOLFOX
Number analyzed (Participants) | 42 | 43 | 41
Percentage of participants | 28.6 [15.7 to 44.6] | 48.8 [33.3 to 64.5] | 39.0 [24.2 to 55.5]
Statistical Analysis 1: Comparison: Phase 2: Axitinib + FOLFOX vs Phase 2: Bevacizumab + FOLFOX; One-sided Cochran-Mantel-Haenszel test of treatment stratified by prior adjuvant chemotherapy (yes versus [vs.] no) and prior pelvic irradiation (yes vs. no) was used for the analysis; Test type: Superiority or Other; p = 0.9726, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.585, 95% CI 2-sided [0.332 to 1.031]
Statistical Analysis 2: Comparison: Phase 2: Axitinib + FOLFOX vs Phase 2: Axitinib + Bevacizumab + FOLFOX; One-sided Cochran-Mantel-Haenszel test of treatment stratified by prior adjuvant chemotherapy (yes vs. no) and prior pelvic irradiation (yes vs. no) was used for the analysis; Test type: Superiority or Other; p = 0.8391, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.735, 95% CI 2-sided [0.399 to 1.352]
Statistical Analysis 3: Comparison: Phase 2: Bevacizumab + FOLFOX vs Phase 2: Axitinib + Bevacizumab + FOLFOX; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.8192, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.797, 95% CI 2-sided [0.489 to 1.299]

2. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUClast) For Axitinib: Phase 1
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast). Pharmacokinetic (PK) parameters of axitinib (AG-013736) were combined for Cohorts 1, 2, and 3. AUClast for axitinib in absence of bevacizumab + FOLFOX was estimated from Cycle 1 Day 8 data and in presence of bevacizumab + FOLFOX was estimated from Cycle 2 Day 1 data. Results were normalized to axitinib 5 mg dose.
Time Frame: Predose, 1, 2, 2.5, 4, 6 and 8 hours postdose on Cycle 1 Day 8, Cycle 2 Day 1
Population: PK parameter analysis set included all treated participants who had at least 1 estimated PK parameters of primary interest. PK assessments were done only for cohort 1 to 5, as per planned analysis. Here 'N' (Number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (95% Confidence Interval); unit: nanogram hour per milliliter (ng*hr/mL)
Groups:
- Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3): Bevacizumab 1, 2 or 5 mg/kg intravenous infusion over 90 minutes on Day 1 of each 14-day cycle followed by FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently with oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily starting from Day 3 in Cycle 1 and starting from Day 1 in all subsequent cycles administered following bevacizumab infusion on Day 1. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFIRI (Cohort 4) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 12 | 6 | 6
nanogram hour per milliliter (ng*hr/mL)
  Cycle 1 Day 8 | 119.02 [56.17 to 252.21] | 106.76 [27.27 to 417.89] | 97.05 [49.01 to 192.16]
  Cycle 2 Day 1 | 95.70 [45.16 to 202.80] | 143.68 [36.70 to 562.43] | 117.47 [59.32 to 232.60]

3. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] For Axitinib: Phase 1
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It was obtained from AUC (0 - t) plus AUC (t - ∞). PK parameters of axitinib (AG-013736) were combined for Cohorts 1, 2, and 3. AUC (t - ∞] for axitinib in absence of bevacizumab + FOLFOX was estimated from Cycle 1 Day 8 data and in presence of bevacizumab + FOLFOX was estimated from Cycle 2 Day 1 data. Results were normalized to axitinib 5 mg dose.
Time Frame: Predose, 1, 2, 2.5, 4, 6, 8 hours postdose on Cycle 1 Day 8, Cycle 2 Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFIRI (Cohort 4) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 8 | 4 | 3
ng*hr/mL
  Cycle 1 Day 8 | 190.51 [77.99 to 465.35] | 113.20 [8.89 to 1442.19] | 205.41 [53.61 to 787.01]
  Cycle 2 Day 1 | 224.46 [91.89 to 548.29] | 168.07 [13.19 to 2141.15] | 178.46 [46.58 to 683.73]

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) For Axitinib: Phase 1
Description: PK parameters of axitinib (AG-013736) were combined for Cohorts 1, 2, and 3.Cmax for axitinib (AG-013736) in absence of bevacizumab + FOLFOX was estimated from Cycle 1 Day 8 data and in presence of bevacizumab + FOLFOX was estimated from Cycle 2 Day 1 data. Results were normalized to axitinib 5 mg dose.
Time Frame: Predose, 1, 2, 2.5, 4, 6, 8 hours postdose on Cycle 1 Day 8, Cycle 2 Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFIRI (Cohort 4) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 12 | 6 | 6
ng/mL
  Cycle 1 Day 8 | 35.57 [18.37 to 68.89] | 27.14 [7.40 to 99.49] | 24.23 [14.32 to 40.98]
  Cycle 2 Day 1 | 27.51 [14.20 to 53.28] | 42.48 [11.59 to 155.73] | 32.62 [19.29 to 55.18]

5. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) For Axitinib: Phase 1
Time Frame: Predose, 1, 2, 2.5, 4, 6, 8 hours postdose on Cycle 1 Day 8, Cycle 2 Day 1
Population: PK assessments were done only for cohort 1 to 5, as per planned analysis. Results for Cmin are not reported because Cmin could not be assessed from the data obtained from the study.
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFIRI (Cohort 4) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Apparent Oral Clearance (CL/F) For Axitinib: Phase 1
Description: Clearance (CL) of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed (F). Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. PK parameters of axitinib (AG-013736) were combined for Cohorts 1, 2, and 3. CL/F for axitinib (AG-013736) in absence of bevacizumab + FOLFOX was estimated from Cycle 1 Day 8 data and in presence of bevacizumab + FOLFOX was estimated from Cycle 2 Day 1 data.
Time Frame: Predose, 1, 2, 2.5, 4, 6, 8 hours postdose on Cycle 1 Day 8, Cycle 2 Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Liter per hour (L/hr)
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFIRI (Cohort 4) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 8 | 4 | 3
Liter per hour (L/hr)
  Cycle 1 Day 8 | 30.01 [15.05 to 59.82] | 47.10 [3.72 to 596.29] | 28.49 [9.32 to 87.03]
  Cycle 2 Day 1 | 30.08 [15.09 to 59.96] | 33.33 [2.63 to 421.92] | 28.90 [9.46 to 88.31]

7. Secondary Outcome: Plasma Decay Half-Life (t1/2) For Axitinib: Phase 1
Description: Plasma decay half-life (t1/2) is the time measured for the plasma concentration to decrease by one half. PK parameters of axitinib (AG-013736) were combined for Cohorts 1, 2, and 3. t1/2 for axitinib in absence of bevacizumab + FOLFOX was estimated from Cycle 1 Day 8 data and in presence of bevacizumab + FOLFOX was estimated from Cycle 2 Day 1 data.
Time Frame: Predose, 1, 2, 2.5, 4, 6, 8 hours postdose on Cycle 1 Day 8, Cycle 2 Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3): Bevacizumab 1,2 or 5 mg/kg intravenous infusion over 90 minutes on Day 1 of each 14-day cycle followed by FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently with oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily starting from Day 3 in Cycle 1 and starting from Day 1 in all subsequent cycles administered following bevacizumab infusion on Day 1. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFIRI (Cohort 4) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 8 | 4 | 3
hours
  Cycle 1 Day 8 | 3.26 (3.943) | 2.23 (0.702) | 3.47 (2.820)
  Cycle 2 Day 1 | 6.12 (7.450) | 3.09 (0.889) | 1.73 (0.456)

8. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUClast) For Oxaliplatin: Phase 1
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast). PK parameters of oxaliplatin, assessed by estimating total platinum in plasma ultrafiltrate, were combined for Cohorts 1, 2, and 3. AUClast for oxaliplatin in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data. Results were normalized to Cycle 1 Day 1 oxaliplatin dose.
Time Frame: Predose, 1, 2, 2.25, 2.5, 4, 6, 8, 24, 36-48 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 15 | 5
ng*hr/mL
  Cycle 1 Day 1 | 4814.87 [4079.46 to 5682.84] | 4308.71 [2822.77 to 6576.87]
  Cycle 2 Day 1 | 5231.71 [4432.64 to 6174.83] | 5303.66 [3474.59 to 8095.57]

9. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] For Oxaliplatin: Phase 1
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It was obtained from AUC (0 - t) plus AUC (t - ∞). PK parameters of oxaliplatin, assessed by estimating total platinum in plasma ultrafiltrate, were combined for Cohorts 1, 2, and 3. AUC (0 - ∞) for oxaliplatin in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data. Results were normalized to Cycle 1 Day 1 oxaliplatin dose.
Time Frame: Predose, 1, 2, 2.25, 2.5, 4, 6, 8, 24, 36-48 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 15 | 5
ng*hr/mL
  Cycle 1 Day 1 | 5955.70 [4615.41 to 7685.21] | 5137.31 [3296.14 to 8006.93]
  Cycle 2 Day 1 | 6744.06 [5226.35 to 8702.50] | 6430.67 [4125.97 to 10022.74]

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) For Oxaliplatin: Phase 1
Description: PK parameters of oxaliplatin, assessed by estimating total platinum in plasma ultrafiltrate, were combined for Cohorts 1, 2, and 3. Cmax for oxaliplatin in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data. Results were normalized to Cycle 1 Day 1 oxaliplatin dose.
Time Frame: Predose, 1, 2, 2.25, 2.5, 4, 6, 8, 24, 36-48 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 15 | 5
ng/mL
  Cycle 1 Day 1 | 278.81 [201.38 to 386.03] | 265.05 [67.62 to 1038.93]
  Cycle 2 Day 1 | 318.99 [230.40 to 441.66] | 374.03 [95.42 to 1466.10]

11. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) For Oxaliplatin: Phase 1
Time Frame: Predose, 1, 2, 2.25, 2.5, 4, 6, 8, 24, 36-48 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 5
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Clearance (CL) For Oxaliplatin: Phase 1
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body. PK parameters of oxaliplatin, assessed by estimating total platinum in plasma ultrafiltrate, were combined for Cohorts 1, 2, and 3. CL for oxaliplatin in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data.
Time Frame: Predose, 1, 2, 2.25, 2.5, 4, 6, 8, 24, 36-48 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: L/hr
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 15 | 5
L/hr
  Cycle 1 Day 1 | 27.51 [21.56 to 35.11] | 30.74 [18.48 to 51.13]
  Cycle 2 Day 1 | 24.29 [19.04 to 31.00] | 24.56 [14.76 to 40.85]

13. Secondary Outcome: Plasma Decay Half-Life (t1/2) For Oxaliplatin: Phase 1
Description: Plasma decay half-life (t1/2) is the time measured for the plasma concentration to decrease by one half. PK parameters of oxaliplatin, assessed by estimating total platinum in plasma ultrafiltrate, were combined for Cohorts 1, 2, and 3. t1/2 for oxaliplatin in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data.
Time Frame: Predose, 1, 2, 2.25, 2.5, 4, 6, 8, 24, 36-48 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 15 | 5
hours
  Cycle 1 Day 1 | 20.63 (6.513) | 18.38 (3.004)
  Cycle 2 Day 1 | 23.30 (14.975) | 19.86 (4.110)

14. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUClast) For 5-Fluorouracil: Phase 1
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast). PK parameters of 5-FU were combined for Cohorts 1, 2, and 3. AUClast for 5-FU in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data. Results were normalized to Cycle 1 Day 1 5-FU dose.
Time Frame: Pre-5-FU bolus, 5 min (post-5-FU bolus), 0.25, 0.5, 0.75, 2, 4, 6, 22, 34-46 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFIRI (Cohort 4) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 14 | 7 | 5
ng*hr/mL
  Cycle 1 Day 1 | 39212.03 [22388.50 to 68677.39] | 40955.29 [23831.07 to 70384.39] | 52164.28 [4725.16 to 575877.57]
  Cycle 2 Day 1 | 45087.71 [25743.27 to 78968.27] | 36533.84 [21258.32 to 62785.83] | 95123.13 [8616.47 to 1050129.94]

15. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] For 5-Fluorouracil: Phase 1
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It was obtained from AUC (0 - t) plus AUC (t - ∞). PK parameters of 5-FU were combined for Cohorts 1, 2, and 3. AUC (0 - ∞) for 5-FU in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data. Results were normalized to Cycle 1 Day 1 5-FU dose.
Time Frame: as for outcome 14
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFIRI (Cohort 4) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 9 | 7 | 5
ng*hr/mL
  Cycle 1 Day 1 | 36314.14 [19623.50 to 67200.90] | 41460.50 [23968.34 to 71718.51] | 52430.15 [4751.38 to 578551.86]
  Cycle 2 Day 1 | 38983.80 [21066.13 to 72141.23] | 36776.79 [21260.68 to 63616.60] | 96632.41 [8757.13 to 1066311.16]

16. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) For 5-Fluorouracil: Phase 1
Description: PK parameters of 5-FU were combined for Cohorts 1, 2, and 3. Cmax for 5-FU in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data. Results were normalized to Cycle 1 Day 1 5-FU dose.
Time Frame: as for outcome 14
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFIRI (Cohort 4) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 14 | 7 | 5
ng/mL
  Cycle 1 Day 1 | 16160.85 [6975.82 to 37439.78] | 34436.94 [22763.46 to 52096.78] | 19622.74 [2754.12 to 139809.41]
  Cycle 2 Day 1 | 16249.77 [7014.20 to 37645.79] | 39730.46 [26262.58 to 60104.90] | 34180.87 [4797.41 to 243534.09]

17. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) For 5-Fluorouracil: Phase 1
Time Frame: Pre-5-FU bolus, 5 min (post-5-FU bolus), 0.25, 0.5, 0.75, 2, 4, 6, 22, 34-48 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 5
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFIRI (Cohort 4) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: Clearance (CL) For 5-Fluorouracil: Phase 1
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body. PK parameters of 5-FU were combined for Cohorts 1, 2, and 3. CL for 5-FU in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data.
Time Frame: as for outcome 14
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: L/hr
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFIRI (Cohort 4) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 9 | 7 | 5
L/hr
  Cycle 1 Day 1 | 147.43 [77.38 to 280.93] | 128.28 [73.44 to 224.05] | 99.36 [10.18 to 969.40]
  Cycle 2 Day 1 | 137.34 [72.08 to 261.70] | 144.62 [82.80 to 252.59] | 53.92 [5.53 to 526.06]

19. Secondary Outcome: Plasma Decay Half-Life (t1/2) For 5-Fluorouracil: Phase 1
Description: Plasma decay half-life (t1/2) is the time measured for the plasma concentration to decrease by one half. PK parameters of 5-FU were combined for Cohorts 1, 2, and 3. t1/2 for 5-FU in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data.
Time Frame: as for outcome 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3) | Phase 1: Axitinib + FOLFIRI (Cohort 4) | Phase 1: Axitinib + FOLFOX (Cohort 5)
Number analyzed (Participants) | 9 | 7 | 5
hours
  Cycle 1 Day 1 | 0.26 (0.218) | 0.19 (0.069) | 0.39 (0.291)
  Cycle 2 Day 1 | 0.25 (0.142) | 0.14 (0.029) | 0.24 (0.131)

20. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUClast) For Irinotecan: Phase 1
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast). AUClast for irinotecan in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data. Results were normalized to Cycle 1 Day 1 irinotecan dose.
Time Frame: Predose, 1, 2, 2.5, 4, 6, 8, 24 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Phase 1: Axitinib + FOLFIRI (Cohort 4)
Number analyzed (Participants) | 7
ng*hr/mL
  Cycle 1 Day 1 | 12081.58 [8805.17 to 16577.15]
  Cycle 2 Day 1 | 11496.32 [8378.62 to 15774.11]

21. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] For Irinotecan: Phase 1
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It was obtained from AUC (0 - t) plus AUC (t - ∞). AUC (0 - ∞) for irinotecan in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data. Results were normalized to Cycle 1 Day 1 irinotecan dose.
Time Frame: Predose, 1, 2, 2.5, 4, 6, 8, 24 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Phase 1: Axitinib + FOLFIRI (Cohort 4)
Number analyzed (Participants) | 7
ng*hr/mL
  Cycle 1 Day 1 | 13055.88 [9371.39 to 18188.96]
  Cycle 2 Day 1 | 12459.89 [8943.60 to 17358.66]

22. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) For Irinotecan: Phase 1
Description: Cmax for irinotecan in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data. Results were normalized to Cycle 1 Day 1 irinotecan dose.
Time Frame: Predose, 1, 2, 2.5, 4, 6, 8, 24 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Phase 1: Axitinib + FOLFIRI (Cohort 4)
Number analyzed (Participants) | 7
ng/mL
  Cycle 1 Day 1 | 1910.25 [1561.45 to 2336.97]
  Cycle 2 Day 1 | 1788.69 [1462.08 to 2188.26]

23. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) For Irinotecan: Phase 1
Time Frame: Predose, 1, 2, 2.5, 4, 6, 8, 24 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 5
Arm/Group | Phase 1: Axitinib + FOLFIRI (Cohort 4)
Number analyzed (Participants) | 0

24. Secondary Outcome: Clearance (CL) For Irinotecan: Phase 1
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body. CL for irinotecan in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data.
Time Frame: Predose, 1, 2, 2.5, 4, 6, 8, 24 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: L/hr
Arm/Group | Phase 1: Axitinib + FOLFIRI (Cohort 4)
Number analyzed (Participants) | 7
L/hr
  Cycle 1 Day 8 | 26.09 [18.10 to 37.61]
  Cycle 2 Day 1 | 27.34 [18.97 to 39.40]

25. Secondary Outcome: Plasma Decay Half-Life (t1/2) For Irinotecan: Phase 1
Description: Plasma decay half-life (t1/2) is the time measured for the plasma concentration to decrease by one half. t1/2 for irinotecan in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data.
Time Frame: Predose, 1, 2, 2.5, 4, 6, 8, 24 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 1: Axitinib + FOLFIRI (Cohort 4)
Number analyzed (Participants) | 7
hours
  Cycle 1 Day 1 | 6.45 (1.406)
  Cycle 2 Day 1 | 6.75 (0.886)

26. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUClast) For Bevacizumab: Phase 1
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast). PK parameters of bevacizumab were combined for Cohorts 1, 2, and 3. AUClast for bevacizumab in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data. The bevacizumab pharmacokinetic parameters were normalized to 1 mg/kg dose.
Time Frame: Predose, 1, 2, 2.25, 2.5, 4, 6, 8, 24, 36-48 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3)
Number analyzed (Participants) | 9
ng*hr/mL
  Cycle 1 Day 1 | 3394758.83 [2453600.72 to 4696928.65]
  Cycle 2 Day 1 | 3554899.52 [2569344.23 to 4918496.49]

27. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] For Bevacizumab: Phase 1
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It was obtained from AUC (0 - t) plus AUC (t - ∞). PK parameters of bevacizumab were combined for Cohorts 1, 2, and 3. AUC (0 - ∞) for bevacizumab in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data. The bevacizumab pharmacokinetic parameters were normalized to 1 mg/kg dose.
Time Frame: Predose, 1, 2, 2.25, 2.5, 4, 6, 8, 24, 36-48 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3)
Number analyzed (Participants) | 9
ng*hr/mL
  Cycle 1 Day 1 | 4987528.96 [3395240.62 to 7326563.24]
  Cycle 2 Day 1 | 5114888.84 [3481940.36 to 7513651.92]

28. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) For Bevacizumab: Phase 1
Description: PK parameters of bevacizumab were combined for Cohorts 1, 2, and 3. Cmax for bevacizumab in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data. The bevacizumab pharmacokinetic parameters were normalized to 1 mg/kg dose.
Time Frame: Predose, 1, 2, 2.25, 2.5, 4, 6, 8, 24, 36-48 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3)
Number analyzed (Participants) | 9
ng/mL
  Cycle 1 Day 1 | 26460.05 [19574.60 to 35767.50]
  Cycle 2 Day 1 | 26850.12 [19863.16 to 36294.76]

29. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) For Bevacizumab: Phase 1
Time Frame: Predose, 1, 2, 2.25, 2.5, 4, 6, 8, 24, 36-48 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 5
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3)
Number analyzed (Participants) | 0

30. Secondary Outcome: Clearance (CL) For Bevacizumab: Phase 1
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body. PK parameters of bevacizumab were combined for Cohorts 1, 2, and 3. CL for bevacizumab in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data.
Time Frame: Predose, 1, 2, 2.25, 2.5, 4, 6, 8, 24, 36-48 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: L/hr
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3)
Number analyzed (Participants) | 9
L/hr
  Cycle 1 Day 1 | 0.01 [0.01 to 0.02]
  Cycle 2 Day 1 | 0.02 [0.01 to 0.02]

31. Secondary Outcome: Plasma Decay Half-Life (t1/2) For Bevacizumab: Phase 1
Description: Plasma decay half-life (t1/2) is the time measured for the plasma concentration to decrease by one half. PK parameters of bevacizumab were combined for Cohorts 1, 2, and 3. t1/2 for bevacizumab in absence of axitinib was estimated from Cycle 1 Day 1 data and in presence of axitinib was estimated from Cycle 2 Day 1 data.
Time Frame: Predose, 1, 2, 2.25, 2.5, 4, 6, 8, 24, 36-48 hours postdose on Cycle 1 Day 1, Cycle 2 Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 1: Axitinib + Bevacizumab + FOLFOX (Cohort 1-3)
Number analyzed (Participants) | 9
hours
  Cycle 1 Day 1 | 205.97 (46.454)
  Cycle 2 Day 1 | 210.22 (55.317)

32. Secondary Outcome: Duration of Response (DR): Phase 2
Description: Time in days from the first documentation of objective tumor response to objective tumor progression or death due to any cancer. Duration of tumor response was calculated as the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1. DR was calculated for the subgroup of participants with a confirmed objective tumor response. CR: disappearance of all lesions and no appearance of new lesions. PR: >=30% decrease in sum of LD of target lesions taking as reference the baseline sum LD, without progression of nontarget lesions and no appearance of new lesions. Progression: >=20% increase in sum of LD of target lesions taking as references the smallest sum LD recorded since treatment start, unequivocal progression of existing nontarget lesions, or appearance of new lesions, occurrence of pleural effusion/ascites, substantiated by cytologic investigation.
Time Frame: as for outcome 1
Population: ITT population included all randomized participants, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug from that to which they were randomized. 'N' (Number of participants analyzed)= those participants who were evaluable for this measure.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Phase 2: Axitinib + FOLFOX: FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently or followed by oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily in each 14-day cycle administered prior to oxaliplatin infusion on Day 1. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 2: Bevacizumab + FOLFOX: Bevacizumab 5 mg/kg intravenous infusion over 90 minutes on Day 1 of each 14-day cycle followed by FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently or followed by oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 2: Axitinib + Bevacizumab + FOLFOX: Bevacizumab 2 mg/kg intravenous infusion over 90 minutes on Day 1 of each 14-day cycle followed by FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently or followed by oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily in each 14-day cycle administered following bevacizumab infusion on Day 1. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
Arm/Group | Phase 2: Axitinib + FOLFOX | Phase 2: Bevacizumab + FOLFOX | Phase 2: Axitinib + Bevacizumab + FOLFOX
Number analyzed (Participants) | 12 | 21 | 16
days | 434.0 [246.0 to 666.0] | NA [232.0 to NA] — Data was not estimable since high number of participants was censored for this measure. | 343.0 [168.0 to 490.0]

33. Secondary Outcome: Progression-Free Survival (PFS): Phase 2
Description: Time in days from date of randomization to first documentation of objective tumor progression or death due to any cause. PFS was calculated as first event date minus the date of first dose of study medication plus 1. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death"). Progression: >=20% increase in sum of LD of target lesions taking as references the smallest sum LD recorded since treatment start, unequivocal progression of existing nontarget lesions, or appearance of new lesions, occurrence of pleural effusion/ascites, substantiated by cytologic investigation.
Time Frame: as for outcome 1
Population: ITT population included all randomized participants, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2: Axitinib + FOLFOX | Phase 2: Bevacizumab + FOLFOX | Phase 2: Axitinib + Bevacizumab + FOLFOX
Number analyzed (Participants) | 42 | 43 | 41
days | 336 [225.0 to 749.0] | 485 [276.0 to NA] — Data was not estimable since high number of participants was censored for this measure. | 381 [238.0 to 425.0]
Statistical Analysis 1: Comparison: Phase 2: Axitinib + FOLFOX vs Phase 2: Bevacizumab + FOLFOX; Hazard ratio and corresponding 95% confidence interval (CI) was calculated based on the Cox proportional hazards model stratified by prior adjuvant chemotherapy (yes vs. no) and prior pelvic irradiation (yes vs. no). One-sided p-value was derived from the log-rank test stratified by prior adjuvant chemotherapy (yes vs. no) and prior pelvic irradiation (yes vs. no); Test type: Superiority or Other; p = 0.5699, Log Rank; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.47 to 2.45]
Statistical Analysis 2: Comparison: Phase 2: Axitinib + FOLFOX vs Phase 2: Axitinib + Bevacizumab + FOLFOX; Hazard ratio and corresponding 95% CI was calculated based on the Cox proportional hazards model stratified by prior adjuvant chemotherapy (yes vs. no) and prior pelvic irradiation (yes vs. no). One-sided p-value was derived from the log-rank test stratified by prior adjuvant chemotherapy (yes vs. no) and prior pelvic irradiation (yes vs. no); Test type: Superiority or Other; p = 0.2167, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.33 to 1.61]
Statistical Analysis 3: Comparison: Phase 2: Bevacizumab + FOLFOX vs Phase 2: Axitinib + Bevacizumab + FOLFOX; [analysis description as in outcome 33, analysis 2]; Test type: Superiority or Other; p = 0.8746, Log Rank; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [0.75 to 2.98]

34. Secondary Outcome: Time to Treatment Failure (TTF): Phase 2
Description: TTF is defined as the time from the randomization to the date of the first documentation of PD, symptomatic deterioration, death due to any cause, or treatment discontinuation due to adverse event, refusal or other reasons. Progression: >=20% increase in sum of LD of target lesions taking as references the smallest sum LD recorded since treatment start, unequivocal progression of existing nontarget lesions, or appearance of new lesions, occurrence of pleural effusion/ascites, substantiated by cytologic investigation.
Time Frame: as for outcome 1
Population: as for outcome 33
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2: Axitinib + FOLFOX | Phase 2: Bevacizumab + FOLFOX | Phase 2: Axitinib + Bevacizumab + FOLFOX
Number analyzed (Participants) | 42 | 43 | 41
days | 187.0 [162.0 to 315.0] | 241.0 [205.0 to 344.0] | 238.0 [155.0 to 333.0]
Statistical Analysis 1: Comparison: Phase 2: Axitinib + FOLFOX vs Phase 2: Bevacizumab + FOLFOX; [analysis description as in outcome 33, analysis 2]; Test type: Superiority or Other; p = 0.8884, Log Rank; Hazard Ratio (HR) = 1.40, 95% CI 2-sided [0.81 to 2.41]
Statistical Analysis 2: Comparison: Phase 2: Axitinib + FOLFOX vs Phase 2: Axitinib + Bevacizumab + FOLFOX; [analysis description as in outcome 33, analysis 2]; Test type: Superiority or Other; p = 0.6648, Log Rank; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.66 to 1.89]
Statistical Analysis 3: Comparison: Phase 2: Bevacizumab + FOLFOX vs Phase 2: Axitinib + Bevacizumab + FOLFOX; [analysis description as in outcome 33, analysis 2]; Test type: Superiority or Other; p = 0.8065, Log Rank; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.75 to 2.07]

35. Secondary Outcome: Overall Survival (OS): Phase 2
Description: Time in days from randomization date to date of death due to any cause. OS was calculated as the death date minus the date of first dose of study medication plus 1. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Every 3 months after discontinuation of study treatment until death due to any cause or 1 year after randomization of the last participant
Population: ITT population included all randomized participants , with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 2: Axitinib + FOLFOX | Phase 2: Bevacizumab + FOLFOX | Phase 2: Axitinib + Bevacizumab + FOLFOX
Number analyzed (Participants) | 42 | 43 | 41
days | 552.0 [443.0 to 911.0] | 659.0 [493.0 to 899.0] | 601.0 [533.0 to 882.0]
Statistical Analysis 1: Comparison: Phase 2: Axitinib + FOLFOX vs Phase 2: Bevacizumab + FOLFOX; [analysis description as in outcome 33, analysis 2]; Test type: Superiority or Other; p = 0.6904, Log Rank; Hazard Ratio (HR) = 1.155, 95% CI 2-sided [0.656 to 2.033]
Statistical Analysis 2: Comparison: Phase 2: Axitinib + FOLFOX vs Phase 2: Axitinib + Bevacizumab + FOLFOX; [analysis description as in outcome 33, analysis 2]; Test type: Superiority or Other; p = 0.7364, Log Rank; Hazard Ratio (HR) = 1.203, 95% CI 2-sided [0.676 to 2.141]
Statistical Analysis 3: Comparison: Phase 2: Bevacizumab + FOLFOX vs Phase 2: Axitinib + Bevacizumab + FOLFOX; [analysis description as in outcome 33, analysis 2]; Test type: Superiority or Other; p = 0.4140, Log Rank; Hazard Ratio (HR) = 0.941, 95% CI 2-sided [0.535 to 1.653]

36. Secondary Outcome: Change From Baseline in M.D. Anderson Symptom Assessment Inventory - Diarrhea (MDASI-D) Symptom Severity and Interference Subscale Scores at Day 1 of Cycle 2 Through Day 1 Cycle 42 and Follow-up: Phase 2
Description: PROs included assessment of symptom severity and interference which were measured using M.D. Anderson Symptom Assessment Inventory-Diarrhea (MDASI-D), 20-item questionnaire which assesses the severity of 14 symptoms over the past 24 hours, as well as symptoms interference with 6 areas of function (e.g., walking, work, mood), when the symptom was "at its worst". Each item is scored from 0 to 10, with '0' indicating that the symptom was either not present or did not interfere with their activities, and '10' indicating that the symptom was "as bad as you can imagine" or "interfered completely" with their life. The 2 subscales, symptom severity score and symptom interference score were average of respective items and ranged from 0 to 10, higher score indicating greater severity or interference of symptoms.
Time Frame: Cycle 1 Day 1 (baseline), every 2 weeks for the first 2 months (Cycle 2 Day 1 [C2D1], Cycle 3 Day 1, and Cycle 4 Day 1) then monthly thereafter starting Cycle 6 Day 1, and 28 days after the last dose
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Phase 2: Axitinib + FOLFOX | Phase 2: Bevacizumab + FOLFOX | Phase 2: Axitinib + Bevacizumab + FOLFOX
Number analyzed (Participants) | 42 | 43 | 41
units on scale
  Severity Scale: Baseline (n=41,43,40) | 1.62 (1.57) | 2.20 (1.93) | 2.18 (2.06)
  Severity Scale: C2D1 (n=37,37,37) | 0.63 (1.22) | 0.04 (1.16) | 0.80 (1.32)
  Severity Scale: C3D1 (n=32,38,32) | 0.68 (1.29) | -0.22 (1.17) | 0.63 (1.61)
  Severity Scale: C4D1 (n=23,37,30) | 0.88 (1.41) | -0.40 (1.27) | 0.64 (1.68)
  Severity Scale: C5D1 (n=23,34,29) | 0.72 (1.37) | -0.34 (1.59) | 0.60 (2.13)
  Severity Scale: C6D1 (n=15,38,26) | 0.70 (1.80) | 0.09 (1.44) | 0.96 (1.60)
  Severity Scale: C7D1 (n=12,30,22) | 0.28 (1.51) | -0.16 (1.55) | 0.26 (1.22)
  Severity Scale: C8D1 (n=17,29,22) | 0.28 (1.45) | -0.13 (1.56) | 0.42 (1.74)
  Severity Scale: C9D1 (n=11,24,21) | -0.15 (1.55) | -0.03 (1.67) | 0.76 (1.50)
  Severity Scale: C10D1 (n=14,27,21) | 0.28 (1.37) | 0.06 (1.52) | 0.77 (1.52)
  Severity Scale: C11D1 (n=10,20,19) | 0.15 (1.57) | -0.05 (1.59) | 0.57 (1.33)
  Severity Scale: C12D1 (n=11,23,16) | 0.32 (1.40) | 0.47 (1.37) | 0.38 (1.14)
  Severity Scale: C13D1 (n=8,13,12) | -0.09 (1.43) | 0.10 (1.35) | 0.73 (1.55)
  Severity Scale: C14D1 (n=8,17,14) | 0.03 (0.81) | 0.38 (1.48) | -0.05 (1.44)
  Severity Scale: C15D1 (n=7,11,9) | 0.28 (1.50) | 0.42 (1.49) | 0.71 (1.34)
  Severity Scale: C16D1 (n=7,17,14) | -0.30 (0.88) | 0.11 (1.46) | 0.05 (2.08)
  Severity Scale: C17D1 (n=5,11,6) | -0.20 (0.70) | 0.21 (1.69) | 0.72 (1.07)
  Severity Scale: C18D1 (n=6,14,9) | 0.02 (0.85) | 0.31 (1.15) | 0.61 (1.55)
  Severity Scale: C19D1 (n=4,8,16) | -0.18 (0.54) | 0.34 (1.42) | 0.81 (2.32)
  Severity Scale: C20D1 (n=5,14,8) | -0.06 (0.54) | 0.15 (1.21) | -0.06 (1.67)
  Severity Scale: C21D1 (n=4,5,5) | -0.25 (0.71) | 0.27 (1.90) | 1.20 (1.35)
  Severity Scale: C22D1 (n=3,11,8) | 0.57 (0.45) | 0.81 (0.95) | 0.09 (1.37)
  Severity Scale: C23D1 (n=4,5,3) | 0.30 (0.80) | 0.64 (1.32) | 1.05 (1.11)
  Severity Scale: C24D1 (n=5,11,7) | 0.91 (2.07) | 0.37 (1.10) | -0.20 (1.62)
  Severity Scale: C25D1 (n=4,5,5) | 0.25 (0.96) | -0.03 (1.12) | -0.30 (1.63)
  Severity Scale: C26D1 (n=4,6,7) | -0.05 (0.76) | 0.46 (0.72) | -0.13 (1.79)
  Severity Scale: C27D1 (n=4,3,4) | -0.21 (0.65) | 0.07 (0.99) | 0.34 (2.70)
  Severity Scale: C28D1 (n=4,5,7) | 0.12 (0.82) | 0.74 (1.01) | -0.43 (2.00)
  Severity Scale: C29D1 (n=2,3,4) | 3.00 (2.12) | -0.14 (0.58) | -0.09 (2.51)
  Severity Scale: C30D1 (n=3,6,3) | 1.05 (1.70) | 0.45 (1.05) | 0.64 (0.68)
  Severity Scale: C31D1 (n=1,1,3) | -0.50 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -0.64 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 1.55 (1.69)
  Severity Scale: C32D1 (n=2,4,4) | 0.11 (0.25) | 0.80 (0.93) | 1.29 (1.03)
  Severity Scale: C33D1 (n=0,0,2) | NA (NA) — Data was not analyzed as no participants were evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable. | 0.89 (1.26)
  Severity Scale: C34D1 (n=2,4,3) | 0.04 (0.15) | 0.75 (0.89) | 0.43 (0.74)
  Severity Scale: C35D1 (n=0,0,1) | NA (NA) — Data was not analyzed as no participants were evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable. | 0.79 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Severity Scale: C36D1 (n=2,3,2) | 0.29 (0.51) | 1.24 (1.22) | -0.18 (0.25)
  Severity Scale: C37D1 (n=0,1,0) | NA (NA) — Data was not analyzed as no participants were evaluable. | 0.86 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Severity Scale: C38D1 (n=2,2,1) | 0.13 (0.28) | 1.68 (1.97) | 0.86 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Severity Scale: C39D1 (n=0,1,0) | NA (NA) — Data was not analyzed as no participants were evaluable. | 0.86 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Severity Scale: C40D1 (n=2,2,2) | 0.18 (0.35) | 1.29 (1.11) | 0.43 (0.61)
  Severity Scale: C42D1 (n=2,2,1) | 0.18 (0.35) | 1.25 (1.26) | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Severity Scale: Follow_Up (n=4,15,14) | 1.29 (2.75) | -0.00 (1.66) | 0.29 (1.72)
  Interference Scale: Baseline (n=41,43,40) | 2.50 (2.70) | 2.79 (2.57) | 2.47 (2.66)
  Interference Scale: C2D1 (n=37,37,36) | 0.46 (1.80) | -0.08 (1.74) | 0.78 (2.55)
  Interference Scale: C3D1 (n=31,38,30) | 0.60 (2.37) | -0.57 (1.88) | 1.09 (2.37)
  Interference Scale: C4D1 (n=23,36,30) | 0.92 (2.16) | -0.54 (1.89) | 1.15 (2.37)
  Interference Scale: C5D1 (n=23,34,29) | 0.65 (2.20) | -0.59 (1.98) | 1.19 (2.90)
  Interference Scale: C6D1 (n=15,38,26) | 0.32 (2.01) | -0.18 (2.33) | 0.99 (2.54)
  Interference Scale: C7D1 (n=12,30,22) | 0.43 (1.25) | -0.59 (2.13) | 0.55 (2.05)
  Interference Scale: C8D1 (n=17,29,22) | 0.01 (1.58) | -0.10 (2.00) | 0.48 (1.87)
  Interference Scale: C9D1 (n=11,24,21) | -0.14 (1.08) | -0.39 (2.31) | 0.75 (1.76)
  Interference Scale: C10D1 (n=14,27,21) | -0.18 (1.80) | 0.15 (2.06) | 0.99 (2.12)
  Interference Scale: C11D1 (n=10,20,19) | 0.42 (1.23) | -0.51 (1.75) | 0.84 (2.50)
  Interference Scale: C12D1 (n=10,23,16) | 0.03 (0.78) | 0.17 (2.23) | 0.38 (1.51)
  Interference Scale: C13D1 (n=8,13,12) | -0.50 (1.56) | -0.31 (2.49) | 0.31 (1.70)
  Interference Scale: C14D1 (n=8,17,14) | -0.10 (0.84) | 0.15 (2.57) | 0.29 (2.12)
  Interference Scale: C15D1 (n=7,11,9) | -0.52 (0.85) | 0.27 (1.91) | 0.70 (2.36)
  Interference Scale: C16D1 (n=7,17,14) | -0.02 (0.33) | -0.48 (2.31) | -0.01 (2.38)
  Interference Scale: C17D1 (n=5,11,6) | -0.90 (1.31) | -0.29 (3.16) | 1.17 (1.28)
  Interference Scale: C18D1 (n=6,14,9) | 0.06 (0.34) | 0.04 (2.38) | 1.00 (2.26)
  Interference Scale: C19D1 (n=4,8,6) | 0.04 (0.34) | 0.54 (2.25) | 1.04 (1.84)
  Interference Scale: C20D1 (n=5,14,8) | 0.27 (0.65) | -0.08 (2.34) | 0.35 (2.07)
  Interference Scale: C21D1 (n=4,5,5) | -0.04 (0.86) | -0.97 (3.50) | 1.83 (1.28)
  Interference Scale: C22D1 (n=3,11,8) | 0.44 (0.84) | 0.74 (1.71) | 0.83 (2.05)
  Interference Scale: C23D1 (n=4,5,3) | 0.21 (0.42) | 1.13 (2.58) | 1.28 (1.80)
  Interference Scale: C24D1 (n=5,11,7) | 2.00 (3.25) | 0.30 (2.65) | 0.55 (2.33)
  Interference Scale: C25D1 (n=4,5,5) | 0.00 (0.41) | 0.10 (2.45) | 0.90 (0.88)
  Interference Scale: C26D1 (n=4,6,7) | 0.33 (0.85) | 0.67 (1.80) | 0.33 (2.11)
  Interference Scale: C27D1 (n=4,3,4) | 0.04 (0.52) | 0.11 (1.13) | 1.63 (2.44)
  Interference Scale: C28D1 (n=4,5,7) | 0.71 (1.19) | 0.97 (1.81) | 0.19 (2.40)
  Interference Scale: C29D1 (n=2,3,4) | 3.25 (3.89) | -0.56 (0.96) | 1.33 (2.97)
  Interference Scale: C30D1 (n=3,6,3) | 0.94 (1.49) | 1.08 (2.16) | 1.06 (1.83)
  Interference Scale: C31D1 (n=1,1,3) | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable. | -0.17 (NA) — Standard deviation was not estimable since only one participant was evaluable. | 2.33 (2.08)
  Interference Scale: C32D1 (n=2,4,4) | 0.08 (0.12) | 1.50 (2.26) | 2.17 (1.81)
  Interference Scale: C33D1 (n=0,0,2) | NA (NA) — Data was not analyzed as no participants were evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable. | 1.92 (2.71)
  Interference Scale: C34D1 (n=2,4,3) | 0.17 (0.24) | 1.25 (1.89) | 1.11 (1.51)
  Interference Scale: C35D1 (n=0,0,1) | NA (NA) — Data was not analyzed as no participants were evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable. | 1.67 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Interference Scale: C36D1 (n=2,3,2) | 0.17 (0.24) | 1.89 (2.18) | 1.33 (1.89)
  Interference Scale: C37D1 (n=0,1,0) | NA (NA) — Data was not analyzed as no participants were evaluable. | 0.83 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Interference Scale: C38D1 (n=2,2,1) | 0.08 (0.12) | 2.25 (2.47) | -0.17 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Interference Scale: C39D1 (n=0,1,0) | NA (NA) — Data was not analyzed as no participants were evaluable. | 0.50 (NA) — Standard deviation was not estimable since only one participant was evaluable. | NA (NA) — Data was not analyzed as no participants were evaluable.
  Interference Scale: C40D1 (n=2,2,2) | 0.42 (0.59) | 2.50 (2.12) | 0.25 (0.35)
  Interference Scale: C42D1 (n=2,2,1) | 0.25 (0.35) | 2.58 (2.24) | 0.00 (NA) — Standard deviation was not estimable since only one participant was evaluable.
  Interference Scale: Follow Up (n=4,15,14) | 1.33 (2.48) | -0.21 (2.44) | 0.91 (1.65)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Phase 1: Axitinib + FOLFOX + Bevacizumab (Cohort 1): Bevacizumab 1 mg/kg intravenous infusion over 90 minutes on Day 1 of each 14-day cycle followed by FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently or followed by oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily starting from Day 3 in Cycle 1 and starting from Day 1 in all subsequent cycles administered following bevacizumab infusion on Day 1. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 1: Axitinib + FOLFOX + Bevacizumab (Cohort 2): Bevacizumab 2 mg/kg intravenous infusion over 90 minutes on Day 1 of each 14-day cycle followed by FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently or followed by oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily starting from Day 3 in Cycle 1 and starting from Day 1 in all subsequent cycles administered following bevacizumab infusion on Day 1. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 1: Axitinib + FOLFOX + Bevacizumab (Cohort 3): Bevacizumab 5 mg/kg intravenous infusion over 90 minutes on Day 1 of each 14-day cycle followed by FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently or followed by oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily starting from Day 3 in Cycle 1 and starting from Day 1 in all subsequent cycles administered following bevacizumab infusion on Day 1. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 1: Axitinib + FOLFIRI (Cohort 4): FOLFIRI combination chemotherapy on Day 1 of each 14-day cycle consisting of irinotecan 180 mg/m^2 intravenous infusion over 90 minutes, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently or followed by irinotecan, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily starting from Day 3 in Cycle 1 and starting from Day 1 in all subsequent cycles administered prior to irinotecan infusion on Day 1. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 1: Axitinib + FOLFOX (Cohort 5): FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently or followed by oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily starting from Day 3 in Cycle 1 and starting from Day 1 in all subsequent cycles administered prior to oxaliplatin infusion on Day 1. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 1: Axitinib + FOLFIRI (Cohort 6): FOLFIRI combination chemotherapy on Day 1 of each 14-day cycle consisting of irinotecan 180 mg/m^2 intravenous infusion over 90 minutes, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently or followed by irinotecan, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily from Day 3 to Day 12 in each 14-day cycle administered following completion of 5-FU infusion on Day 3. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 1: Axitinib + FOLFOX (Cohort 7): FOLFOX combination chemotherapy on Day 1 of each 14-day cycle consisting of oxaliplatin 85 mg/m^2 intravenous infusion over 2 hours, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently or followed by oxaliplatin, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 5 mg orally twice daily starting from Day 3 to Day 12 in each 14-day cycle administered following completion of 5-FU infusion on Day 3. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 1: Axitinib + FOLFIRI (Cohort 8): Axitinib (AG-13736) tablet 7 mg orally twice daily for 7 days in 2-week lead-in period prior to Day 1 Cycle 1. FOLFIRI combination chemotherapy on Day 1 of each 14-day cycle consisting of irinotecan 180 mg/m^2 intravenous infusion over 90 minutes, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently or followed by irinotecan, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 7 mg to 10 mg orally twice daily from Day 3 to Day 9 in each 14-day cycle administered following completion of 5-FU infusion on Day 3. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
- Phase 1: Axitinib + FOLFOX (Cohort 9): Axitinib (AG-13736) tablet 7 mg orally twice daily for 7 days in 2-week lead-in period prior to Day 1 Cycle 1. FOLFIRI combination chemotherapy on Day 1 of each 14-day cycle consisting of irinotecan 180 mg/m^2 intravenous infusion over 90 minutes, leucovorin 400 mg/m^2 intravenous infusion over 2 hours administered concurrently or followed by irinotecan, then 5-FU 400 mg/m^2 intravenous bolus injection and a subsequent 5-FU 2400 mg/m^2 intravenous infusion over 46 to 48 hours. Axitinib (AG-013736) tablet 10 mg orally twice daily from Day 3 to Day 9 in each 14-day cycle administered following completion of 5-FU infusion on Day 3. Dose adjustment for any drug in the combination was done for individual participants who experienced drug-related toxicity, as per investigator's discretion.
Arm/Group | Phase 1: Axitinib + FOLFOX + Bevacizumab (Cohort 1) | Phase 1: Axitinib + FOLFOX + Bevacizumab (Cohort 2) | Phase 1: Axitinib + FOLFOX + Bevacizumab (Cohort 3) | Phase 1: Axitinib + FOLFIRI (Cohort 4) | Phase 1: Axitinib + FOLFOX (Cohort 5) | Phase 1: Axitinib + FOLFIRI (Cohort 6) | Phase 1: Axitinib + FOLFOX (Cohort 7) | Phase 1: Axitinib + FOLFIRI (Cohort 8) | Phase 1: Axitinib + FOLFOX (Cohort 9) | Phase 2: Axitinib + FOLFOX | Phase 2: Bevacizumab + FOLFOX | Phase 2: Axitinib + Bevacizumab + FOLFOX
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/6 | 2/4 | 3/8 | 5/6 | 1/4 | 1/6 | 1/3 | 8/18 | 15/39 | 17/43 | 23/41
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 4/4 | 8/8 | 6/6 | 4/4 | 6/6 | 3/3 | 18/18 | 39/39 | 42/43 | 39/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Axitinib + FOLFOX + Bevacizumab (Cohort 1) (N=6) | Phase 1: Axitinib + FOLFOX + Bevacizumab (Cohort 2) (N=6) | Phase 1: Axitinib + FOLFOX + Bevacizumab (Cohort 3) (N=4) | Phase 1: Axitinib + FOLFIRI (Cohort 4) (N=8) | Phase 1: Axitinib + FOLFOX (Cohort 5) (N=6) | Phase 1: Axitinib + FOLFIRI (Cohort 6) (N=4) | Phase 1: Axitinib + FOLFOX (Cohort 7) (N=6) | Phase 1: Axitinib + FOLFIRI (Cohort 8) (N=3) | Phase 1: Axitinib + FOLFOX (Cohort 9) (N=18) | Phase 2: Axitinib + FOLFOX (N=39) | Phase 2: Bevacizumab + FOLFOX (N=43) | Phase 2: Axitinib + Bevacizumab + FOLFOX (N=41)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gastrointestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Sepsis syndrome (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 2 | 7
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aortic thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Axitinib + FOLFOX + Bevacizumab (Cohort 1) (N=6) | Phase 1: Axitinib + FOLFOX + Bevacizumab (Cohort 2) (N=6) | Phase 1: Axitinib + FOLFOX + Bevacizumab (Cohort 3) (N=4) | Phase 1: Axitinib + FOLFIRI (Cohort 4) (N=8) | Phase 1: Axitinib + FOLFOX (Cohort 5) (N=6) | Phase 1: Axitinib + FOLFIRI (Cohort 6) (N=4) | Phase 1: Axitinib + FOLFOX (Cohort 7) (N=6) | Phase 1: Axitinib + FOLFIRI (Cohort 8) (N=3) | Phase 1: Axitinib + FOLFOX (Cohort 9) (N=18) | Phase 2: Axitinib + FOLFOX (N=39) | Phase 2: Bevacizumab + FOLFOX (N=43) | Phase 2: Axitinib + Bevacizumab + FOLFOX (N=41)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 1 | 2 | 3 | 1 | 1 | 5 | 9 | 9 | 12
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 4 | 2 | 3 | 3
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Microcytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 3 | 1 | 1 | 1 | 2 | 9 | 15 | 21 | 19
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 2 | 2 | 1 | 1 | 0 | 6 | 11 | 12 | 16
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3 | 1 | 2
Deafness (Ear and labyrinth disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 2 | 2 | 3 | 7 | 2 | 7
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 3 | 3 | 2 | 0 | 1 | 0 | 5 | 8 | 5 | 14
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 12
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 4
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 3 | 1 | 3
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 4 | 3 | 5 | 5 | 3 | 5 | 3 | 13 | 22 | 23 | 23
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 4 | 7
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 7
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 2 | 4 | 5 | 9
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 1 | 5 | 0 | 1 | 2 | 3 | 6 | 12 | 12 | 15
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Asthenia (General disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 1 | 8 | 5 | 4
Axillary pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site haematoma (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 3
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4
Chills (General disorders) | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 3 | 1 | 2
Device dislocation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device occlusion (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 4 | 4 | 4 | 3 | 4 | 4 | 2 | 14 | 24 | 29 | 31
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hernia pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 4
Mucosal inflammation (General disorders) | 6 | 2 | 1 | 2 | 4 | 2 | 1 | 1 | 6 | 7 | 9 | 15
Nodule (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 4 | 5 | 4 | 3
Pain (General disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 6 | 4
Pyrexia (General disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 4 | 3 | 6 | 8
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 10 | 9
Thrombosis in device (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Arthropod-borne disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 5
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Enterobacter sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Incision site infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 3
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 2 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinea infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 4 | 3
Urinary tract infection (Infections and infestations) | 3 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 3 | 5 | 3 | 7
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound dehiscence (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure diastolic decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1
Blood testosterone decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 1
Cardiac enzymes increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 2 | 1 | 2 | 1 | 0 | 1 | 2 | 2 | 7 | 6 | 17
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 4 | 2 | 4 | 4 | 0 | 3 | 1 | 5 | 10 | 10 | 20
Dehydration (Metabolism and nutrition disorders) | 5 | 0 | 0 | 4 | 3 | 0 | 1 | 1 | 3 | 7 | 8 | 12
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 3 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3 | 1 | 1 | 0 | 0 | 5 | 7 | 7 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 4 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 4 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 3 | 4 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 3 | 4 | 6 | 3 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Bursa disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 6 | 0 | 4
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 4 | 4 | 7
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 4
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 2 | 2 | 2 | 0 | 2 | 2 | 3 | 8 | 6 | 7
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 5 | 8
Headache (Nervous system disorders) | 4 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 5 | 8 | 6 | 13
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1
IIIrd nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Mononeuritis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 2 | 4 | 0 | 2 | 0 | 4 | 0 | 5 | 12 | 23 | 17
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 5 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 9 | 6 | 8
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 4 | 5
Claustrophobia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 5 | 9
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 2 | 2 | 1 | 0 | 0 | 1 | 1 | 11 | 7 | 10
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 3 | 3 | 3
Glycosuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 3 | 5 | 5 | 12
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urge incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 3 | 6 | 7 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 2 | 8 | 1 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 2 | 1 | 1 | 0 | 2 | 6 | 5 | 8 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 4 | 3 | 0 | 2 | 1 | 1 | 10 | 13 | 12
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 3 | 2 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 6
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 2 | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 4 | 4 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 4 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Facial wasting (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 5 | 1 | 7
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Plantar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 3 | 1 | 1 | 0 | 3 | 7 | 3 | 8
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 3
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 6 | 3 | 4 | 2 | 2 | 2 | 2 | 2 | 8 | 16 | 8 | 26
Hypotension (Vascular disorders) | 1 | 1 | 0 | 5 | 0 | 0 | 0 | 1 | 6 | 1 | 5 | 7
Intermittent claudication (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2

LIMITATIONS AND CAVEATS:
Time to Treatment Failure (TTF) was included as a secondary endpoint of the study after change in analysis plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.